CLINICAL TRIAL: NCT04854356
Title: The Effects of Blood Flow Restriction During High-intensity Interval Exercise Among Healthy Adult Males: a Randomized Controlled Trial
Brief Title: Blood Flow Restriction During High-intensity Interval Exercise
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universiti Sains Malaysia (Other)
Responsible Party: Principal Investigator, Shazlin Shaharudin, Lecturer, Universiti Sains Malaysia
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: USM/JEPeM/20060331
Record Dates: First submitted 2021-04-15; First posted 2021-04-22 (Actual); Last update posted 2021-04-22 (Actual); Status verified 2021-04

CONDITIONS: Exercise Physiology; Biomechanics
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HIE with BFR during exercise phase (Experimental): BFR with 40% Arterial occlusive pressure cycling at 85% VO2max for 3 minutes and rest interval for 3 minutes (4 sets) each time during exercise
  Interventions: Other: Exercise with blood flow restriction (BFR)
- HIE with BFR during interval phase (Active Comparator): BFR with 40% Arterial occlusive pressure cycling at 85% VO2max for 3 minutes and rest interval for 3 minutes (4 sets) each during the interval
  Interventions: Other: Exercise with blood flow restriction (BFR)
- HIE without BFR (No Intervention): Cycling at 85% VO2max for 3 minutes and rest interval for 3 minutes (4 sets) each time during exercise

INTERVENTIONS:
Other: Exercise with blood flow restriction (BFR) — All participants completed high-intensity interval exercise plus (1) BFR applied during exercise phase, or (2) BFR applied during interval phase, or (3) no BFR applied.
  Arms: HIE with BFR during exercise phase; HIE with BFR during interval phase

SUMMARY:
The study is a randomized controlled trial aimed to compare the effects of blood flow restriction (BFR) in different phases (i.e., exercise versus interval) during high-intensity interval exercise (HIIE) on aerobic capacity, anaerobic capacity, isokinetic knee strength, lower limb biomechanics during single-leg landing and cycling economy among healthy adult males. Participants were randomized to three groups. Intervention was conducted for 12 weeks with 2 sessions per week. During intervention, all groups conducted HIEE on cycle ergometer with or without BFR. Assessments were conducted before the intervention, on the 6th week of intervention and after the intervention. Assessments included physical characteristics, aerobic and anaerobic capacity, lower limb biomechanics during single-leg landing and isokinetic knee strength.

DETAILED DESCRIPTION:
The study is a randomized controlled trial aimed to compare the effects of blood flow restriction (BFR) in different phases (i.e., exercise versus interval) during high-intensity interval exercise on aerobic capacity, anaerobic capacity, isokinetic knee strength, lower limb biomechanics during single-leg landing and cycling economy among healthy adult males. The procedure of the study has been approved by Ethics Committee of Universiti Sains Malaysia (USM/JEPeM/20060331) and complied with the Declaration of Helsinki. participants were randomised into one of the following conditions: 1. High-intensity interval exercise without BFR (C Group). 2. High-intensity interval exercise with BFR during exercise phase (E Group). 3 High-intensity interval exercise with BFR during interval phase (I Group). After obtaining the participants' written informed consent form, participants proceeded to pre-intervention tests. Each exercise test needs to be separated by at least 24 hours (First day: VO2max; Second day: Cycling economy; Third day: Isokinetic knee strength and Wingate tests). In the sixth week and after the twelfth week of the exercise intervention, the participants took part in the mid-test and post-test, which was similar protocol in the pre-test. The duration of the intervention is 12 weeks, with two sessions per week. Each exercise session took about an hour and monitored by an exercise physiologist. Exercise intervention comprised of cycle exercises using a cycle ergometer device. First, participants performed a 5-minute warm-up activity (50W). After the warm-up, each group sprinted with 85% VO2max for 3 minutes, where the rotation speed should be maintained at around 60 revolutions per minute (RPM) and then rests for 3 minutes on the ergometer without cycling. Then, they sprinted again after the first break and this sequence of sprint and rest were repeated three times. The 85% of VO2max was determined based on the results from the VO2max test. Exercise (E) Group and Interval (I) Group completed the training with an air cuff placed at the inguinal fold of both legs in sequence in order to provide partial blood flow restriction. The sequence of wrapping was done in random order, but both thighs were wrapped twice in a single intervention session. E Group applied 40% LOP BFR during exercise; I Group I applied 40% LOP BFR during passive rest i.e., interval. On the other hand, C group does not perform BFR during the whole process. Two-factor repeated measures analysis of variance (pre-, mid-and post-intervention time points x three groups) was used to examine the main effects and interaction effects of changes for each tested variables following intervention. If the main effects or interaction effects are significant, the Newman-Keuls post hoc test was applied for multiple comparisons.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male adults.
2. Age between 20-25.
3. Have normal body mass index (BMI).
4. Physically active (i.e., exercise regularly for at least three times per week) and total score more than 600MET-min/week based on The International Physical Activity Questionnaire (IPAQ).
5. VO2max value above 42 ml/kg/min during cycling test (Above fair VO2max level)(American College of Sports Medicine, 2010).

Exclusion Criteria:

1. BMI is greater than 25kg/m2.
2. Have exercise-related disorders such as coronary heart disease, peripheral vascular diseases, rhabdomyolysis, respiratory inflammation, or have neurological disorders.
3. Have implanted electrical devices.
4. Have significant cognitive impairment.

Ages: 20 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
Change of aerobic capacity from baseline to post-intervention | 12 weeks
  Maximum oxygen consumption was measured during Astrand protocol
Change of anaerobic capacity from baseline to post-intervention | 12 weeks
  Maximum power was measured during Wingate test protocol
Change of muscular strength from baseline to post-intervention | 12 weeks
  The strength of the thigh muscle groups was measured using isokinetic device
Change of knee joint moments from baseline to post-intervention | 12 weeks
  Biomechanical data measured during single-leg landing test

CONTACTS AND LOCATIONS:
Overall Officials: Shazlin Shaharudin, Principal Investigator — Universiti Sains Malaysia
Locations (1):
- Universiti Sains Malaysia, Kota Bharu, Kelantan, Malaysia

IPD SHARING:
Plan to Share IPD: No
All data in the experiment is anonymous and has been stored in SPSS software. Only researchers can view or extract data. Data were shown as grouped data and participants were not individually identified. The data must be password protected, and only the researcher can access all the data. Before taking the photos and wearing a gas collection mask, the researcher had to ask the participants' permission. The three-dimensional video recorded using Qualisys could not identify the respondent as it only captured the reflective marker number's trajectory on the respondent. Data will be published as scientific articles to be shared with other researchers.